CLINICAL TRIAL: NCT01322763
Title: Prevalence of Sleep Apnea/Hypopnea Syndrome in Obese Children. The Significance of Hormonal Factors
Brief Title: Prevalence of Sleep Apnea/Hypopnea Syndrome in Obese Children
Acronym: NANOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Juan Ruiz Manzano, Spanish Society of Pneumology and Thoracic Surgery
Other Study IDs: PI755
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Sleep Apnea; Children; Obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Principal aim: To determine the prevalence of Sleep Apnea- Hypopnea syndrome in obese children.

Secondary aim: 1. To fix the implication of the adenotonsillar hypertrophy, the obesity and the hormonal factors in the pathogeny of SAHS in children. 2. To determinate of clinical and neurophysiologic characteristics of childhood SAHS associated with obesity. DESIGN: A prospective transversal study.

DETAILED DESCRIPTION:
The population of study will be make for children of both sex, between 3 and 14 years old and with body mass index (BMI) ≥ 95 percentile and with informed consent. METHODS: In all children included in the study, the investigators will carry out: previous history, history of snoring and Chervin´s screening questionnaire of SAHS, general physical and otorhinolaryngologic examination with nasopharyngoscopy, blood test with determination of glucose, lipids, insulin, leptin, adiponectin, and ghrelin, polysomnography (PSG) with transcutaneous CO2. The diagnosis of SAHS will be made if on PSG the Respiratory disturbance Index (RDI) is ≥ 3 and/or obstructive hypoventilation is present.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sex, between 3 and 14 years old
* Body mass index (BMI) ≥ 95 percentile
* With informed consent.

Exclusion Criteria:

* Without informed consent

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population of study will be make for children of both sex, between 3 and 14 years old and with body mass index (BMI) ≥ 95 percentile and with informed consent.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-05 (Estimated); Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luz Alonso-Álvarez, MD, Principal Investigator — Sleep Unit. Complejo Asistencial Universitario Burgos. Spain
Locations (1):
- Complejo Asistencial Universitario de Burgos, Burgos, Burgos, Spain

REFERENCES:
- [Derived] Alonso-Alvarez ML, Teran-Santos J, Gonzalez Martinez M, Cordero-Guevara JA, Jurado-Luque MJ, Corral-Penafiel J, Duran-Cantolla J, Ordax Carbajo E, MasaJimenez F, Kheirandish-Gozal L, Gozal D; Spanish Sleep Network. Metabolic biomarkers in community obese children: effect of obstructive sleep apnea and its treatment. Sleep Med. 2017 Sep;37:1-9. doi: 10.1016/j.sleep.2017.06.002. Epub 2017 Jun 22. PMID 28899517
- [Derived] Alonso-Alvarez ML, Teran-Santos J, Navazo-Eguia AI, Martinez MG, Jurado-Luque MJ, Corral-Penafiel J, Duran-Cantolla J, Cordero-Guevara JA, Kheirandish-Gozal L, Gozal D; Spanish Sleep Network. Treatment outcomes of obstructive sleep apnoea in obese community-dwelling children: the NANOS study. Eur Respir J. 2015 Sep;46(3):717-27. doi: 10.1183/09031936.00013815. Epub 2015 Jun 11. PMID 26065566
- [Derived] Kheirandish-Gozal L, Gileles-Hillel A, Alonso-Alvarez ML, Peris E, Bhattacharjee R, Teran-Santos J, Duran-Cantolla J, Gozal D. Effects of adenotonsillectomy on plasma inflammatory biomarkers in obese children with obstructive sleep apnea: A community-based study. Int J Obes (Lond). 2015 Jul;39(7):1094-100. doi: 10.1038/ijo.2015.37. Epub 2015 Mar 24. PMID 25801692
- [Derived] Gileles-Hillel A, Alonso-Alvarez ML, Kheirandish-Gozal L, Peris E, Cordero-Guevara JA, Teran-Santos J, Martinez MG, Jurado-Luque MJ, Corral-Penafiel J, Duran-Cantolla J, Gozal D. Inflammatory markers and obstructive sleep apnea in obese children: the NANOS study. Mediators Inflamm. 2014;2014:605280. doi: 10.1155/2014/605280. Epub 2014 Jun 1. PMID 24991089
- [Derived] Alonso-Alvarez ML, Cordero-Guevara JA, Teran-Santos J, Gonzalez-Martinez M, Jurado-Luque MJ, Corral-Penafiel J, Duran-Cantolla J, Kheirandish-Gozal L, Gozal D. Obstructive sleep apnea in obese community-dwelling children: the NANOS study. Sleep. 2014 May 1;37(5):943-9. doi: 10.5665/sleep.3666. PMID 24790273